CLINICAL TRIAL: NCT01459510
Title: A Brief Multimedia Program Affects Parents' Attitudes Toward Physical Punishment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 100533
Record Dates: First submitted 2011-07-25; First posted 2011-10-25 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Violence Prevention
Keywords: Violence prevention; Parenting; Discipline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- multi media intervention (Experimental): Play Nicely Program
  Interventions: Behavioral: Play Nicely Program
- Routine primary care (No Intervention): Routine primary care

INTERVENTIONS:
Behavioral: Play Nicely Program — Multi media educational intervention
  Arms: multi media intervention

SUMMARY:
The American Academy of Pediatrics recommends that parents receive anticipatory guidance about how to discipline their children as part of the well child visit. However, physicians provide counseling only 25-40% of the time. In regard to the type of discipline, the AAP recommends that primary care providers encourage parent to use non-physical forms of discipline and discourage parents from using physical punishment. Educational resources are needed to help physicians routinely provide these important anticipatory guidance messages. In this study, consecutive parents were exposed to routine anticipatory guidance messages before the well child visit with the physician. After the clinic visit, parents were invited to participate in a research study to assess their attitudes about physical punishment and other discipline strategies. The key research question of this study is: Can a brief multimedia program (i.e. Play Nicely program) affect parents' attitudes about the use of physical punishment? The time frame of the study was June through August of 2010. Data was collected immediately after the clinic visit and 2-4 weeks post clinic visit.

DETAILED DESCRIPTION:
Note: Because of a poor follow up rate with the 2-4 week phone call, this effort to collect follow up data was unsuccessful.

ELIGIBILITY:
English and Spanish speaking parents of 6-24 month old children presenting for a primary care visit in the Vanderbilt Pediatric Primary Care Clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Attitudes toward spanking | Immediately post clinic visit
  After the clinic visit, parents were invited to participate in a 2 minute survey which included the ATS scale, a 10 item scale that is associated with parents' actual use of physical punishment. Data was obtained from the parent immediately after the clinic visit while the parent was in the clinic. We attempted a follow up phone call 2-4 weeks post clinic visit. However, due to a poor follow up rate, this data will not be reported nor will it be compared to the data that was collected immediately post clinic visit.

CONTACTS AND LOCATIONS:
Overall Officials: Seth J Scholer, MD, MPH, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Medical Center, Primary clinic, Nashville, Tennessee, United States

REFERENCES:
- [Background] Scholer SJ, Hamilton EC, Johnson MC, Scott TA. A brief intervention may affect parents' attitudes toward using less physical punishment. Fam Community Health. 2010 Apr-Jun;33(2):106-16. doi: 10.1097/FCH.0b013e3181d592ef. PMID 20216353
- [Background] Scholer SJ, Hudnut-Beumler J, Dietrich MS. A brief primary care intervention helps parents develop plans to discipline. Pediatrics. 2010 Feb;125(2):e242-9. doi: 10.1542/peds.2009-0874. Epub 2010 Jan 18. PMID 20083523
- [Derived] Chavis A, Hudnut-Beumler J, Webb MW, Neely JA, Bickman L, Dietrich MS, Scholer SJ. A brief intervention affects parents' attitudes toward using less physical punishment. Child Abuse Negl. 2013 Dec;37(12):1192-201. doi: 10.1016/j.chiabu.2013.06.003. Epub 2013 Jul 13. PMID 23859768
- See also: Website for program that teaches discipline strategies — http://www.playnicely.org